CLINICAL TRIAL: NCT01087346
Title: Mothers' Thoughts About What Their Children Eat
Brief Title: Mothers' Thoughts About Kids and Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 100076; 10-HG-0076
Record Dates: First submitted 2010-03-13; First posted 2010-03-16 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Overweight
Keywords: Risk Perception; Obesity Risk; Healthy Volunteer; HV
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Active Comparator): Information about child health
  Interventions: Behavioral: Reading Information
- Family Environment Information (Experimental): Information about family environment factors in children's obesity risk
  Interventions: Behavioral: Reading Information
- Gene times Family Environment Information (Experimental): Information about interactions between genetic and family environment factors in children's obesity risk
  Interventions: Behavioral: Reading Information
- Genetic Information (Experimental): Information about genetic factors in child obesity risk
  Interventions: Behavioral: Reading Information

INTERVENTIONS:
Behavioral: Reading Information — Reading information about risk factors for obesity among children

SUMMARY:
Summary:

* A few studies have explored the effects of providing parents with health information about their children. However, more information is needed about the relationship between awareness of health information and changes in behavior. This study will investigate the impact of health information on choices that parents make about food for their children.
* Mothers and fathers with a biological child between the ages of 3-7 years old may be eligible for this study. Participants are recruited from the Washington, DC metropolitan area.
* In this study, before visiting the research center, participants will answer online questionnaires about their children's health and eating habits and their own health and eating habits.
* At the research center, participants will use a virtual reality model of a buffet to make food choices for their children. Participants will be introduced to the computer-based virtual buffet scenario as a training session to prepare for using the buffet during the experimental context. While in the virtual environment, participants wear a virtual reality helmet that allows them to see the virtual buffet scenario.
* After the training session, participants will watch an interactive computer presentation about a health topic.
* Participants will then visit the virtual buffet scenario again for the formal session, and will choose a virtual lunch meal for their child as before.
* At the end of their visit, participants will complete post-test questionnaires about their experiences during the experiment and other research-related information.
* Participants will be asked to complete a follow-up questionnaire online a week after their visit
* The total time for the study visit is approximately 90 minutes. The participants children will not be asked to take part in the study.

Eligibility:

- Men and Women at least 18 years of age who have a biological child between the ages of 3 and 7 who has no major diet-related health conditions, developmental delays, or disabilities. You may not take part in the study if you have a history of seizures and/or are pregnant.

DETAILED DESCRIPTION:
Purpose

This study will investigate the impact of health information on choices that parents make about food for their children. Participants will use a virtual reality model of a buffet to make food choices.

Mothers and fathers with a biological child between the ages of 3-7 years old may be eligible for this study. Participants are recruited from the Washington, DC metropolitan area.

Study participants will complete THREE sets of surveys and one task. Participants will complete a web-based survey before coming in for a study appointment. When participants arrive for their appointment, they will watch an interactive presentation on health information. Next, participants will interact in a virtual reality environment and will be asked to select virtual lunch for their child from a buffet. While in the virtual environment, a participant wears a head-mounted virtual reality headset that allows him/her to see elements of the environment. Participants will complete an additional computer-based survey. Finally, participants will be asked to complete an online questionnaire a week following their visit. The total time for the study visit is approximately 90 minutes. The participants children will not be asked to take part in the study.

Detailed Description

This study will investigate issues around the impact of health information on choices that parents make about food for their children. Participants will perform tasks that include completing computer-based surveys, watching an interactive computer-based presentation about health information, participating in a virtual reality model by selecting virtual lunch for their children from a buffet, and completing a computed-based exit survey. As part of the study, participants will wear a virtual reality helmet and be immersed in a buffet where they will select virtual lunch for their child.

For this study, we are only recruiting men and women that have a biological child between the ages of 3-7 years old. You may not take part in the study if you have a history of seizures and/or are pregnant.

ELIGIBILITY:
* INCLUSION CRITERIA :

Study 1:

All participants will be healthy adult women over the age of 18 (though in practice the age range is likely to be constrained naturally by the required age of the index child).

1. having a self-reported body mass index of greater than or equal to 25
2. having some amount of familiarity with their family health history
3. having a biological child between the ages of 4 and 5 inclusive, who lives in the same household at least 1 day out of the past 30 days, and who has no major food allergies or diet-related health conditions, developmental delays, or disabilities
4. having the ability to read and write in English
5. being able to come to the NIH Clinical Center for one visit

EXCLUSION CRITERIA:

1. having a vestibular or seizure disorder;
2. having a high propensity for motion sickness;
3. known pregnancy; (4) uncorrected low vision or hearing;

(5) inability to complete tasks in the virtual environment;

(6) past or current history of eating disorder;

(7) NHGRI employees

Study 2:

INCLUSION CRITERIA:

All participants will be healthy adults over the age of 18 (though in practice the age range is likely to be constrained naturally by the required age of the index child).

1. having a self-perception of being overweight
2. having a biological child between the ages of 3 and 7

   inclusive (of any weight), who has no food allergies to buffet items (e.g., dairy, wheat, fruit) or diet-related health conditions, developmental delays, or disabilities that would severely limit food

   choices on the virtual buffet and who does not have a vegan or gluten-free diet
3. self-reporting that the parent is responsible for feeding to the child to criterion
4. having the ability to read and write in English
5. being able to come to the NIH Clinical Center for one visit

EXCLUSION CRITERIA:

1. having a vestibular or seizure disorder
2. having a high propensity for motion sickness
3. known pregnancy
4. uncorrected low vision or hearing
5. inability to complete tasks in the virtual environment
6. past or current history of eating disorder
7. NHGRI employees
8. having another household member or another biological parent of their index child having participated in the study
9. women who report being pregnant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1148 (Actual)
Dates: Start 2010-11-19 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
The number of calories selected for participant's index child in a virtual buffet food selection task | 1 visit
  The number of calories selected for participant's index child in a virtual buffet food selection task

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Persky, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Bouhlal S, Abrams LR, McBride CM, Persky S. Cognitive and affective factors linking mothers' perceived weight history to child feeding. Eur J Clin Nutr. 2018 Nov;72(11):1583-1591. doi: 10.1038/s41430-017-0071-0. Epub 2018 Feb 6. PMID 29410480
- [Derived] Bouhlal S, McBride CM, Ward DS, Persky S. Drivers of overweight mothers' food choice behaviors depend on child gender. Appetite. 2015 Jan;84:154-60. doi: 10.1016/j.appet.2014.09.024. Epub 2014 Oct 6. PMID 25300916
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-HG-0076.html